CLINICAL TRIAL: NCT01434615
Title: SASHFR (South Asian Systolic Heart Failure Registry) : A Multi-center, Nonrandomized, Prospective Study to Collect Data Pertaining to the Demographic and Cardiovascular Profiles, Management Strategies and Clinical Outcomes of HF Patients.
Brief Title: Medtronic South Asian Systolic Heart Failure Registry
Acronym: SASHFR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SASHFR; CTRI/2008/091/000203 (Registry Identifier: Clinical Trials Registry - India)
Record Dates: First submitted 2011-09-13; First posted 2011-09-15 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Heart Failure
Keywords: Cardiac Resynchronization Therapy; Moderate to advanced; patients; current consensus guidelines
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No-CRT (Experimental): Patients who meet CRT device implantation guidelines (i.e., meet CRT indication and on optimal medical therapy) but who do not get a CRT-P or CRT-D device implanted
  Interventions: Other: No-CRT
- CRT (Experimental): Patients who meet CRT device implantation guidelines (i.e., meet CRT indication and on optimal medical therapy) and receive CRT-P or CRT-D device
  Interventions: Device: CRT

INTERVENTIONS:
Device: CRT — Patients who meet CRT device implantation guidelines (i.e., meet CRT indication and on optimal medical therapy) and receive CRT-P or CRT-D device
  Arms: CRT
Other: No-CRT — Patients who meet CRT device implantation guidelines (i.e., meet CRT indication and on optimal medical therapy) but who do not get a CRT-P or CRT-D device implanted
  Arms: No-CRT

SUMMARY:
The purpose of this study is to (a) characterize the current management of patients with systolic heart failure (HF) in South Asia following an educational intervention of current guidelines and delivery of disease management tools and (b) to characterize the effect of current therapy on clinical outcomes in patients managed by tertiary care centers across South Asia. Current therapy includes characterization of the post market performance of any market released Medtronic cardiac resynchronization therapy (CRT) or cardiac resynchronization therapy plus implantable cardiac defibrillator (CRT-D) system for cardiac resynchronization therapy (CRT).

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed and dated study informed consent. Patients having moderate to severe heart failure (NYHA Class III or IV) EF < 35% as measured by echo, MUGA, contrast ventriculogram or MRI. QRS duration > 120 ms.

Exclusion Criteria:

Patient has life expectancy of less than 12 months due to medical conditions other than HF.

* Patient has experienced unstable angina, acute myocardial infarction (MI), coronary artery bypass graft (CABG) or percutaneous transluminal coronary angioplasty (PTCA) within the past 3 months.
* Patient is known to have chronic permanent atrial arrhythmias (i.e., cases of long-standing atrial fibrillation of greater than 1 year, including those in which cardioversion has not been indicated or attempted).
* Patient is enrolled in any concurrent study that would confound the results of this study.
* Patient is pregnant or breastfeeding.
* Patient has a CRT device implanted previously.
* Patient has had a heart transplant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Clinical Composite score | 2 years
  1. To characterize the long term outcomes (clinical composite score as improved, unchanged or worsened) of patients who meet CRT implant guidelines and (a) receive CRT implant or (b) do not receive the CRT implant.

SECONDARY OUTCOMES:
Demographics | 2 years FU
  To determine the demographics of HF patients in the registry including LVEF and NYHA Classification.
Profile of patients with positive response to CRT | 2 years
  To characterize the profile of patients with a positive response to CRT. e.g Baseline LVEF

CONTACTS AND LOCATIONS:
Overall Officials: C Narasimhan, Principal Investigator — Care Hospital, Hyderabd-India
Locations (1):
- Care Hospital, Hyderabad, Andhra Pradesh, India